CLINICAL TRIAL: NCT02982044
Title: Endothelial Function Responses to Manipulations in Blood Flow Pattern
Brief Title: Artery Function Responses to Changes in Blood Flow
Acronym: ASPEN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Natural Sciences and Engineering Research Council, Canada (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ASPEN
Record Dates: First submitted 2016-11-24; First posted 2016-12-05 (Estimated); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Endothelial Dysfunction
Keywords: blood flow; endothelial function; shear stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Experimental-Control (Experimental): Participants will undergo all interventions, while simultaneously serving as their own within-subject control. The left side of the body will be designated "experimental", and all interventions will be applied to the left arm. The right side of the body will be designated as "control", and will not receive any interventions.
  Interventions: Other: Suprasystolic (300 mmHg) cuff compressions; Other: Handgrip exercise; Other: Passive heat stress

INTERVENTIONS:
Other: Suprasystolic (300 mmHg) cuff compressions — 10 minutes of ECG-gated repeated suprasystolic (300 mmHg) cuff compressions, with inflation occurring every other heart cycle. These cuff compressions may be triggered 0 seconds, 0.2 seconds, or 0.4 seconds from the R spike (systole) on the ECG signal.
Other: Handgrip exercise — 10 minutes of ECG-gated rhythmic handgrip exercise at 30% maximal voluntary contraction, with contraction occurring every other heart cycle
Other: Passive heat stress — 10 minutes of passive heat stress at 42 degrees Celsius with a commercially available heating blanket

SUMMARY:
The purpose of this study is to determine if different blood flow patterns change artery function. We hypothesize that the temporary induction of an oscillatory blood flow pattern will result in an immediate improvement in artery function. Participants will be asked to come to the Vascular Dynamics Lab (IWC E102) at McMaster University for a total of 3 visits. The first visit will allow the participant to get comfortable with the lab and the upcoming tests; and the next 2 visits will be scheduled at the same time of day to collect data. For visits 2 and 3, participants will be asked to arrive after a 4 hour fast. At these visits, ultrasound imaging will be used to examine the arteries and how they may change when blood flow patterns through an artery in the arm are changed. To change blood flow in the arm, heat, rhythmic squeezing of the forearm with a cuff, or handgrip exercise will be used. These interventions will be applied to the left forearm, from the elbow to the fingertips. A trained technician will also draw a blood sample during both data collection visits. A total of 10 participants will be recruited for the entire study.

DETAILED DESCRIPTION:
Interested individuals will be invited to the lab for a screening and familiarization visit, in which the brachial artery (BA) will be scanned to vet for image quality and a BA flow-mediated dilation test will be performed to ensure participant tolerance during collection visits. All qualified participants will be instructed to refrain from vigorous physical activity > 24 hours, alcohol and caffeine > 6 hours, and food > 4 hours prior to each of the two collection visits. Upon arrival, basic anthropometric measures will be collected and hematocrit will be measured in duplicate with a finger prick blood sample equivalent to two 70 µl capillary tubes. Each of the two data collection visits will begin 10 minutes of supine rest, while the participant is instrumented with skin temperature probes on the forearms and hands for measurement of skin temperature, single-lead ECG (Powerlab model ML795, ADInstruments, Colorado Springs, CO, USA) and non-invasive finger cuff (Finometer MIDI, Finapres, The Netherlands) for continuous heart rate and blood pressure monitoring. On the first data collection visit, following rest, the participant will then undergo three 10-minute interventions applied to the left forearm in the following sequence: (1) ECG-gated suprasystolic (300 mmHg) cuff compressions with inflation occurring every other heart cycle, (2) 42 °C heating with a heating blanket, and (3) ECG-gated rhythmic handgrip exercise at 30% MVC with contraction occurring every other heart cycle. 10-minute rest periods will separate each of the interventions to allow for return to baseline conditions. On the second data collection visit, following rest, the participant will undergo three variations of the 10-minute cuff compression intervention, the order of which will be randomized. The three variations differ in the trigger delay from the R spike of the ECG to cause inflation of the cuff for compressions. The original intervention involves the data acquisition unit triggering inflation of the cuff at systole (R spike) (0s delay). This condition will be compared to two other trigger delays, specifically triggering inflation of the cuff at 0.2s and 0.4s after the R spike. For both data collection visits, BA blood velocities, blood flow turbulence, endothelial shear stress, and oscillatory shear index will be assessed before and during each of the interventions; and relative flow-mediated dilation will be assessed before and immediately after each of the interventions. Participants will provide written informed consent prior to beginning any portion of the study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy (no cardiovascular, musculoskeletal, or metabolic disease)
* Male
* 18-35 years old
* Recreationally active (exercising 2-3 times per week)

Exclusion Criteria:

* Cardiovascular, musculoskeletal, or metabolic disease

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Brachial artery flow-mediated dilation | Up to 2 weeks
  Collected using vascular ultrasound and analyzed using semi-automated edge-tracking software

SECONDARY OUTCOMES:
Mean blood velocity magnitude and direction | Up to 2 weeks
  Collected using vascular ultrasound and sent to spectral analyzer for calculation of intensity-weighted mean
Reynolds number (blood flow turbulence) | Up to 2 weeks
  Calculated using blood velocity and artery diameter obtained from vascular ultrasound, and blood density and viscosity calculated using hematocrit
Endothelial shear stress | Up to 2 weeks
  Calculated using blood velocity and artery diameter obtained from vascular ultrasound, and blood viscosity calculated using hematocrit
Oscillatory shear index | Up to 2 weeks
  Calculated using blood velocity and artery diameter obtained from vascular ultrasound
Endothelial shear rate | Up to 2 weeks
  Calculated using blood velocity and artery diameter obtained from vascular ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Maureen J MacDonald, PhD, Principal Investigator — McMaster University
Locations (1):
- McMaster University Vascular Dynamics Lab, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang C, Baker BM, Chen CS, Schwartz MA. Endothelial cell sensing of flow direction. Arterioscler Thromb Vasc Biol. 2013 Sep;33(9):2130-6. doi: 10.1161/ATVBAHA.113.301826. Epub 2013 Jun 27. PMID 23814115
- [Background] Tinken TM, Thijssen DH, Hopkins N, Dawson EA, Cable NT, Green DJ. Shear stress mediates endothelial adaptations to exercise training in humans. Hypertension. 2010 Feb;55(2):312-8. doi: 10.1161/HYPERTENSIONAHA.109.146282. Epub 2010 Jan 4. PMID 20048193
- [Background] Thijssen DH, Dawson EA, Black MA, Hopman MT, Cable NT, Green DJ. Brachial artery blood flow responses to different modalities of lower limb exercise. Med Sci Sports Exerc. 2009 May;41(5):1072-9. doi: 10.1249/MSS.0b013e3181923957. PMID 19346980
- [Background] Gurovich AN, Braith RW. Enhanced external counterpulsation creates acute blood flow patterns responsible for improved flow-mediated dilation in humans. Hypertens Res. 2013 Apr;36(4):297-305. doi: 10.1038/hr.2012.169. Epub 2012 Oct 18. PMID 23076403
- [Background] Reneman RS, Arts T, Hoeks AP. Wall shear stress--an important determinant of endothelial cell function and structure--in the arterial system in vivo. Discrepancies with theory. J Vasc Res. 2006;43(3):251-69. doi: 10.1159/000091648. Epub 2006 Feb 20. PMID 16491020
- [Background] Totosy de Zepetnek JO, Ditor DS, Au JS, MacDonald MJ. Impact of shear rate pattern on upper and lower limb conduit artery endothelial function in both spinal cord-injured and able-bodied men. Exp Physiol. 2015 Oct;100(10):1107-17. doi: 10.1113/EP085056. Epub 2015 Aug 18. PMID 26206681